CLINICAL TRIAL: NCT04018014
Title: Low-dose CT Angiography in the Detection of Acute Pulmonary Embolism: Validation in an Obese Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2019 CASSAGNES
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-07

CONDITIONS: Pulmonary Embolism; Obesity; CT Scanner
Keywords: Pulmonary embolism; Obesity; CT scanner; Iterative reconstructions
MeSH Terms: conditions — Pulmonary Embolism; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- < 30 kg/m2: patients with BMI < 30/kg/m2
  Interventions: Other: CT angiography
- >30 kg/m2: patients with BMI > 30 kg/m2
  Interventions: Other: CT angiography

INTERVENTIONS:
Other: CT angiography — CT angiography in detection of pulmonary embolism

SUMMARY:
Pulmonary embolism is a common pathology in the general population, whose suspicion is based on the clinical and dosage of D-dimers in particular.

The key examination for the diagnosis of pulmonary embolism is chest CT angiography (negative predictive value of 98%).

The evolution of machines in recent years allows a reduction of possible kilovoltage up to 80 kV, different computer algorithms (iterative reconstructions) to reconstruct the images and thus reduce the irradiation dose with equal image quality (Evaluation of dose CT and adaptive statistical reconstruction with the same group of patients, Qi et al, 2012; Impact of iterative reconstruction on the diagnosis of acute pulmonary embolism (PE) on reduced-dose chest CT angiograms, Pontana et al , 2015) in patient populations with a weight of less than 100 kilos.

However, obesity is a risk factor for pulmonary embolism and the obese population is increasing, thus requiring optimal management regarding irradiation.

Few studies have evaluated the quality of low dose CT angiography in obese patients. One study showed the possibility of performing low-dose thoracic CT angiography (100 kV) in patients up to 125 kg, without loss of subjective quality (but with an impact on objective quality), without the use of current iterative reconstruction techniques (Diagnostic confidence and image quality of CT pulmonary angiography at 100 kVp in overweight and obese patients, Megyeri et al, 2015).

The study seek to prove that in the obese patient, with a low dose examination (voltage of the tube at 100 kV) and the current iterative reconstructions, the thoracic angioscanner is not less efficient than in the non obese patient, that the qualities objective and subjective analyzes are maintained.

The main purpose is to evaluate and compare thoracic CT angiography with weight and BMI, with identical CT parameters (same voltage, computer reconstruction techniques and same contrast injection protocol), by evaluating the objective and subjective diagnostic quality of the opacification of the pulmonary arteries.

DETAILED DESCRIPTION:
The study is monocentric, realised in University Hospital of Clermont-Ferrand, France, using the CT GE Revolution dedicated to the emergency service.

For each patient with suspicion of pulmonary embolism, regarding the inclusion and exclusion criteria (explained later), investigators realise the same protocol.

Patients are divided into 2 groups of weight : <30 kg/m2, > 30 kg/m2. There is no change in the management of patients, who benefit from an angioscan for pulmonary embolism, with an optimized protocol for patients under 100 kg and validated by the literature (Megyeri et al. , 2015) for patients over 100 kilos, with no loss of diagnostic chance and with an improvement over the irradiation compared to the usual protocols used (over-irradiation in the obese, up to 140 kV).

Concerning the CT protocol, a voltage of 100 kV is applied (irradiation 40% lower than a 120 kV test), with a modulation of the intensity of the current according to the Z axis and use of different levels of iterative reconstructions on images obtained to improve diagnostic performance.

Regarding the injection protocol, the same product with high concentration of iodine is injected to all patients (IOMERON 400), with a quantity relative to the weight of 1 mL / kg of patient weight, a maximum of 90 mL, a rate of 4 mL / s and rinsing with 30 mL of saline solution at 3 mL / sec

The session physician first carries out diagnostic work by searching for pulmonary embolism or an alternative diagnosis to explain the symptoms.

Secondly, the research work is carried out and the analyzed data with evaluation of the objective diagnostic quality, placing regions of circular interest or ROI (for regions of interest), in the pulmonary arteries, up to the sub-segmental branches.

The subjective quality is evaluated by two double-blind readers by a subjective quality scale.

The different elements are then compared according to two different groups of weights and BMIs. Intermediate statistical analyzes are planned for all 30 patients.

The study started on March 21st, for an estimated duration of 6 months initially. 65

ELIGIBILITY:
Inclusion criteria :

* Patient > 18
* Suspicion of pulmonary embolism
* Reparted in 2 groups :
* < 30 kg/m2
* > 30 kg/m2

Exclusion criteria :

* Allergy to iodine contrast media
* Renal impairment with renal creatinine clearance < 30 mL/min
* Pregnancy
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspicion of pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Unit of hounsfield (UH) measurement in region of interest (ROI) | Day 0
  Unit of hounsfield (UH) measurement in region of interest (ROI) in the pulmonary artery, right and left branches, lobar branches, one segmental and subsegmental branch for each lobe, signal / noise ratio and contrast / noise for each ROI

SECONDARY OUTCOMES:
Scale of confidence (Likert) | Day 0
  Scale of confidence (Likert) on the subjective quality for each reader (2 readers) in 5 points : Total confidence, Good confidence, Neither good or bad confidence, Bad confidence, No confidence at all. Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lucie CASSAGNES, MD-PHD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Background] Megyeri B, Christe A, Schindera ST, Horkay E, Sikula J, Cullmann JL, Kollar J, Heverhagen JT, Szucs-Farkas Z. Diagnostic confidence and image quality of CT pulmonary angiography at 100 kVp in overweight and obese patients. Clin Radiol. 2015 Jan;70(1):54-61. doi: 10.1016/j.crad.2014.09.014. Epub 2014 Oct 24. PMID 25459197